CLINICAL TRIAL: NCT01207011
Title: A Randomised, Open-Label Phase 3 Trial Comparing Amrubicin Versus Docetaxel in Patients With Non-Small Cell Lung Cancer After Failure of First-Line Chemotherapy
Brief Title: Amrubicin (AMR) Trial in Patients With Non-small Cell Lung Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sumitomo Pharma Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D0702035
Record Dates: First submitted 2010-09-21; First posted 2010-09-22 (Estimated); Last update posted 2022-04-12 (Actual); Status verified 2022-04

CONDITIONS: Lung Cancer
MeSH Terms: conditions — Lung Neoplasms | interventions — Docetaxel

ARMS (2):
- 1 AMR (Experimental)
  Interventions: Drug: Amrubicin hydrocloride
- 2 DOC (Active Comparator)
  Interventions: Drug: Docetaxel

INTERVENTIONS:
Drug: Amrubicin hydrocloride — AMR was administered i.v. by 35mg/m2 at day 1, 2 and 3 followed by 3 week rest as 1 course.
  Arms: 1 AMR
Drug: Docetaxel — DOC was administered i.v. by 60mg/m2 at day 1 followed by 3 week rest as 1 course.
  Arms: 2 DOC

SUMMARY:
The study is to evaluate the effect of amrubicin (AMR) compared to docetaxel (DOC) in the treatment of non-small cell lung cancer (NSCLC).

ELIGIBILITY:
Inclusion Criteria:

* Histological or cytological diagnosis of non-small cell lung cancer (NSCLC)
* 1 or 2 prior chemotherapy regimen including 1 platinum-based chemotherapy
* 20 or older but younger than 75 years of age

Exclusion Criteria:

* Symptomatic brain metastasis
* Interstitial pneumonia or pulmonary fibrosis
* Abnormal cardiac function or myocardial infraction within 6 months before study enrollment
* Active infection

Ages: 20 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 202 (Actual)
Dates: Start 2010-10; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Progression free survival | 3.3 months

SECONDARY OUTCOMES:
Overall survival | 12 months
response rate (RECIST) | 3 months
Number of Participants with Adverse Events | 4 months

CONTACTS AND LOCATIONS:
Locations (1):
- 32 Sites, Multiple Locations, Japan

REFERENCES:
- [Derived] Yoshioka H, Katakami N, Okamoto H, Iwamoto Y, Seto T, Takahashi T, Sunaga N, Kudoh S, Chikamori K, Harada M, Tanaka H, Saito H, Saka H, Takeda K, Nogami N, Masuda N, Harada T, Kitagawa H, Horio H, Yamanaka T, Fukuoka M, Yamamoto N, Nakagawa K. A randomized, open-label, phase III trial comparing amrubicin versus docetaxel in patients with previously treated non-small-cell lung cancer. Ann Oncol. 2017 Feb 1;28(2):285-291. doi: 10.1093/annonc/mdw621. PMID 28426104